CLINICAL TRIAL: NCT00545298
Title: An Investigation of the Topical Application of Gaseous Nitric Oxide on Safety and Efficacy in Venous Stasis Leg Ulcers of the Lower Extremities
Brief Title: Safety and Efficacy of Gaseous Nitric Oxide on Venous Stasis Leg Ulcers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic direction of the sponsor changed
Sponsor: Nitric BioTherapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP 1
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-10

CONDITIONS: Venous Ulcers
Keywords: Nitric Oxide; Venous Leg Ulcers
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A - Standard of Care (control) (No Intervention): Standard of care - dressings and sustained compression only
- B Same treatment for 6 weeks (Experimental): 200ppm NO gas 8hrs/day 6 weeks NO gas in nitrogen is delivered constantly to a patch over the wound
  Interventions: Drug: Nitric Oxide - same dose 6 wks
- C - modified treatment, 5 wks lower dose (Experimental): 200 ppm No gas 8 hrs/day 1 wk, 20ppm 8hrs/day 5 weeks Gas is NO in nitrogen delivered constantly for 8 hours to a patch over the wound
  Interventions: Drug: Nitric Oxide modified treatment

INTERVENTIONS:
Drug: Nitric Oxide - same dose 6 wks — 200ppm, 8hrs / day for 6 weeks NO gas in nitrogen delivered to a patch over the wound
  Arms: B Same treatment for 6 weeks
Drug: Nitric Oxide modified treatment — 200ppm, 8hrs/day for 1 week, followed by 25ppm 8hrs/day for 5 weeks Gas is delivered to a patch over the wound
  Arms: C - modified treatment, 5 wks lower dose

SUMMARY:
This study will test the safety and efficacy of nitric oxide gas in the treatment of venous leg ulcers

DETAILED DESCRIPTION:
Prospective, single center. Controlled study of a moisture retentive wound dressing and sustained compression with 6 weeks of 8 hour daily nitric oxide treatments.

ELIGIBILITY:
Inclusion Criteria:

* Must have a venous stasis ulcer between the knee and the ankle.
* Ulcer duration must be 60 days or greater

Exclusion Criteria:

* Has an ulcer that is deemed by the Investigator to be caused primarily by a medical condition other than venous insufficiency
* Suffers from diabetes mellitus with HbA1c ≥ 8%
* Suffers from clinically significant arterial disease
* Is pregnant, a nursing mother or a woman of child bearing potential who is not using an adequate form of contraception (or abstinent)

The above is a partial list of the inclusion and exclusion criteria; however, other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph V Boykin, MD, Principal Investigator — HCA Retreat Hospital
Locations (1):
- Retreat Hospital, Wound Healing Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: single site, 4 subjects recruited starting in October, 2007 with the last vist on August 28, 2008
Groups:
- B - Same Treatment for 6 Weeks: 200ppm NO gas 8hrs/day 6 weeks NO gas in nitrogen is delivered constantly to a patch over the wound
Period: Overall Study
Arm/Group | A - Standard of Care (Control) | B - Same Treatment for 6 Weeks | C - Modified Treatment, 5 Wks Lower Dose
Started | 2 | 1 | 1
Completed | 0 | 1 | 0
Not Completed | 2 | 0 | 1
Not completed — Issues with Standard of Care | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Standard of Care (Control) | B Same Treatment for 6 Weeks | C - Modified Treatment, 5 Wks Lower Dose | Total
Number analyzed (Participants) | 2 | 1 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 2
  >=65 years | 2 | 0 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 76 (4) | 60 (0) | 65 (0) | 69 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Wound Healing
Description: % Re-epithelialization
Time Frame: Week 20
Population: Per protocol. Only one subject met the 20 week time point. All other subjects withdrew early from the study and did not reach the Week 20 time point
Measure: Number; unit: % re-epithelialization
Groups:
- B - Same Treatment for 6 Weeks: This group received 200ppm NO in Nitrogen delivered constantly to a patch over the wound for 8 hours per day for 6 weeks
- C - Modified Treatment, 5 Wks Lower Dose: 200 ppm NO gas 8 hrs / day 1 wk, 20ppm 8 hrs / day 5 weeks. Gas is NO in nitrogen delivered constantly for 8 hours to a patch over the wound
Arm/Group | B - Same Treatment for 6 Weeks | A - Standard of Care (Control) | C - Modified Treatment, 5 Wks Lower Dose
Number analyzed (Participants) | 1 | 0 | 0
% re-epithelialization | 10 |  |

2. Primary Outcome: Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: All reported adverse events, related or unrelated to the study drug.
Time Frame: up to 24 weeks
Population: All enrolled subjects, 4 in total
Measure: Number; unit: number of events
Arm/Group | A - Standard of Care (Control) | B - Same Treatment for 6 Weeks | C - Modified Treatment, 5 Wks Lower Dose
Number analyzed (Participants) | 2 | 1 | 1
number of events
  AEs | 4 | 4 | 7
  SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Arm/Group | A - Standard of Care (Control) | B Same Treatment for 6 Weeks | C - Modified Treatment, 5 Wks Lower Dose
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Standard of Care (Control) (N=2) | B Same Treatment for 6 Weeks (N=1) | C - Modified Treatment, 5 Wks Lower Dose (N=1)
Pain/ Compression Wrap (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Paronychia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — paronychia was considered severe
epistaxis (General disorders) | 0 (0) | 1 (2) | 0 (0)
blister formation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
deterioration of the wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (3)
viral illness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
wound infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to small number of subjects enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is only allowed to publish the results of the trial with the permission of the Sponsor